CLINICAL TRIAL: NCT04177251
Title: Cardiovascular Fibrosis in Idiopathic Pulmonary Fibrosis
Acronym: CardioIPF
Status: Completed | Type: Observational
Sponsor: San Gerardo Hospital (Other)
Responsible Party: Principal Investigator, Paola Faverio, Principal Investigator, San Gerardo Hospital
Other Study IDs: 1349/2019
Record Dates: First submitted 2019-11-19; First posted 2019-11-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Idiopathic Pulmonary Fibrosis; Cardiac Fibrosis; Arterial Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples collected at T1 for:
  1. ELISA assay for periostin, galectin n-3, osteopontin and pro-BNP determination
  2. metabolomic and proteomic analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fibroproliferative diseases, including pulmonary, cardiac and vascular fibrosis share common pathogenetic mechanisms. Furthermore, cardiovascular comorbidities are frequently found in patients with IPF. However, the prevalence of cardiac and vascular fibrosis in patients with IPF have yet to be determined.

Main Purpose of this study is to evaluate, with non-invasive methods (echocardiogram, endothelial function and pulse wave velocity) and blood biomarkers (galectins-3, osteopontin, periostin and pro-BNP), the presence of vascular fibrosis (vascular rigidity and endothelial function) and cardiac fibrosis (prevalence of HFpEF - Heart Failure with Preserved Ejection Fraction) in patients with idiopathic pulmonary fibrosis (IPF), compared to healthy controls.

DETAILED DESCRIPTION:
Fibroproliferative diseases are the cause of 45% of deaths in developed countries. A wide range of diseases belongs to this category, including pulmonary fibrosis.

The fact that in some fibroproliferative diseases the fibrotic process may involve several organs suggests the activation of common causative and pathophysiological mechanisms, which involve inflammatory cells - in particular macrophages and T lymphocytes - epithelial and endothelial cells and fibrogenesis effector cells (fibroblasts, myofibroblasts and fibrocytes). Even in fibroproliferative diseases that apparently have no multiorgan manifestations, such as idiopathic pulmonary fibrosis (IPF), idiopathic myelofibrosis and cardiac fibrosis, common pathogenic pathways have already been studied and recognized (e.g. metabolic pathway of the transforming growth factor-beta -TGF-β- and activation of the transcription factor c-JUN which cause uncontrolled production of collagen fibers by fibroblasts).

Furthermore, cardiovascular comorbidities are frequently found in patients with IPF, particularly ischemic heart disease and arrhythmias. With regard to ischemic heart disease the prevalence reported in patients with IPF is directly proportional to the high prevalence of left ventricular diastolic dysfunction. However, the nature of the association between IPF and ischemic heart disease as well as the prevalence of cardiac and vascular fibrosis in patients with IPF have yet to be determined.

The primary purpose of our study is to evaluate, with non-invasive methods (echocardiogram, endothelial function and pulse wave velocity) and blood biomarkers (galectins-3, osteopontin, periostin and pro-BNP), the presence of vascular fibrosis (vascular rigidity and endothelial function) and cardiac fibrosis (prevalence of HFpEF - Heart Failure with Preserved Ejection Fraction) in patients with idiopathic pulmonary fibrosis (IPF), compared to the general population.

Secondary purposes are the evaluation of the association between the presence and the degree of pulmonary-cardiac-vascular fibrosis and the level of biomarkers analysed (pro-BNP, galectins-3, osteopontin and periostin) and the evaluation of the association between the presence / degree of vascular and / or cardiac fibrosis at baseline and disease progression at 1 year from the diagnosis of IPF.

Explorative aim of the study is also to evaluate the association between the degree of pulmonary fibrosis and the levels of blood proteomic and metabolomic biomarkers measured at baseline only in IPF patients.

Study design: multicenter observational case-control study. For IPF patients, participation in the study consists of two visits (T1, at IPF diagnosis, and T3, 1 year after T1) at the IPF clinic where the patient is followed up, as per normal clinical practice. Clinical history, arterial blood gas analysis and / or SpO2, pulmonary function tests and DLco and 6 minutes walking tests will be collected at T1 and T3. Blood samples for pro-BNP, galectin-n3, osteopontin, periostin and proteomic / metabolomic analysis will be collected at T1. A cardiological evaluation (T2), within 1 month of T1, will be performed in order to collect cardiological clinical data and to perform the following non-invasive measurements: echocardiogram, flow mediated dilation (FMD), pulse wave velocity (PWV).

For healthy volunteers the participation in the study consists of a baseline visit during which cardiopulmonary physical examination, clinical data and blood samples for biomarkers will be collected (T1). A cardiological examination with echocardiogram, FMD and PWV will take place within 1 month from T1.

ELIGIBILITY:
For IPF patients:

Inclusion Criteria:

* diagnosis of idiopathic pulmonary fibrosis according to the 2011 ATS / ERS guidelines with Multidisciplinary discussion;
* informed consent signed and obtained before study enrollment.

Exclusion Criteria:

* having already received (currently or in the past) therapy with pirfenidone or nintedanib;
* participation in other experimental interventional protocols with medicinal use;
* need for oxygen therapy at rest;
* active smoking;
* presence of atrial fibrillation or atrial flutter;
* amputation of a limb or severe peripheral vasculopathy (defined as the presence of previous stenting or vascular surgery of the lower limbs or as the presence of claudication with onset of symptoms for intervals <700 m).

For healthy volunteers:

Inclusion Criteria:

- informed consent signed and obtained before study enrollment.

Exclusion Criteria:

* active smoking;
* presence of atrial fibrillation or atrial flutter;
* amputation of a limb or severe peripheral vasculopathy (defined as the presence of previous stenting or vascular surgery of the lower limbs or as the presence of claudication with onset of symptoms for intervals <700 m);
* diagnostic suspicion of IPF at baseline (T1);
* participation in other experimental protocols.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with diagnosis of IPF
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
presence of cardiac fibrosis in a population of patients with overt IPF at diagnosis in comparison with healthy controls | During visit 2 (T2) (to be performed within 1 month from visit 1) - duration 1day
  Cardiac fibrosis will be evaluated with echocardiography and defined according to the latest guidelines on heart failure as the presence of signs and symptoms of cardiac instability (dyspnea on exertion, asthenia, pulmonary or peripheral congestion) with the finding of a conserved EF (> 50%), the presence of high NT-proBNP (> 125 pg / mL) and one of the following two criteria: 1 - presence of left ventricular hypertrophy (septal thickness) > = 11 mm or indexed left ventricular mass> 125 g / m2 in men or> 95 g / m2 in women) or left atrial dilation (area> 20 cm2 or atrial volume> 55 mL); 2 - presence of diastolic dysfunction from 2nd to 4th grade (assessed by the E / A, dec time and E / E 'ratio echocardiography). Given the new definition in the guidelines of heart failure for intermediate EF (equal criteria but with EF between 40 and 49%) this diagnosis will also be taken into account.
presence of vascular fibrosis in a population of patients with overt IPF at diagnosis in comparison with healthy controls | During visit 2 (T2) (to be performed within 1 month from visit 1) - duration 1 day
  Vascular fibrosis is measured with FMD and PWV, a value less than 4% and greater than 10 cm / s, respectively, will be indicative of a reduction in endothelial function and an increase in vascular stiffness. It is sufficient for one of the two parameters to exceed the threshold value in order to diagnose vascular fibrosis.

SECONDARY OUTCOMES:
levels of biomarkers analysed (galectins-3, osteopontin and periostin) | visit 1 (T1) - duration 1 day
  levels of biomarkers analysed will be evaluated through ELISA tests
IPF progression after 1 year from diagnosis in IPF patients | up yo 1 year
  IPF progression is defined as at least one of the following a) absolute decrease of 10% of predicted compared to the baseline in the forced vital capacity (FVC), or b) absolute decrease of 15% of predicted compared to the baseline in the DLco, or c) acute exacerbation of IPF, or d) IPF-related death, or e) lung transplantation, or f) hospitalisation for respiratory causes.

OTHER OUTCOMES:
blood proteomic and metabolomic biomarkers | during visit 1 (T1) - duration 1 day
  proteomic and metabolomic biomarkers will be identified through metabolomic and proteomic analyses

CONTACTS AND LOCATIONS:
Overall Officials: Paola Faverio, MD, Principal Investigator — Università degli Studi di Milano Bicocca - Ospedale San Gerardo
Locations (1):
- Ospedale San Gerardo Monza - Università Milano Bicocca, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: Undecided